CLINICAL TRIAL: NCT00528567
Title: An International Multi-centre Open-label 2-arm Phase III Trial of Adjuvant Bevacizumab in "Triple Negative" Breast Cancer.
Brief Title: BEATRICE Study: A Study of Bevacizumab (Avastin) Adjuvant Therapy in Triple Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20289; 2007-001128-11 (EudraCT Number)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

ARMS (2):
- Bevacizumab and Chemotherapy (Experimental): Participants randomized to receive bevacizumab in combination with chemotherapy as prescribed.
  Interventions: Drug: Bevacizumab; Drug: Standard adjuvant chemotherapy
- Chemotherapy (Active Comparator): Participants randomized to receive standard adjuvant chemotherapy as prescribed.
  Interventions: Drug: Standard adjuvant chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was administered at a dose equivalent of 5 mg/kg/week using 1 of 3 different scheduling options depending on the schedule of the adjuvant chemotherapy regimen selected for an individual patient.
  Other Names: Avastin
  Arms: Bevacizumab and Chemotherapy
Drug: Standard adjuvant chemotherapy — All chemotherapy schedules and doses for each patient were prescribed according to the labeled indication of the country in which the patient was receiving therapy.

SUMMARY:
The main objective of the trial is to compare Invasive Disease-Free Survival (IDFS) of patients randomised to treatment with adjuvant chemotherapy alone or to adjuvant chemotherapy with 1 year of bevacizumab.

The secondary objectives of this trial are to:

* compare Overall Survival (OS), Breast Cancer-Free Interval (BCFI), Disease- Free Survival (DFS) and Distant Disease-Free Survival (DDFS) of patients randomised to treatment with adjuvant chemotherapy alone or to adjuvant chemotherapy in combination with 1 year of bevacizumab
* evaluate the safety and tolerability of bevacizumab

An exploratory sub-study (not reported here) was to identify biomarkers (from tumour or serum) predictive of toxicity and for the level of benefit from the addition of bevacizumab to standard adjuvant systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* operable primary invasive breast cancer;
* completed definitive loco-regional surgery;
* primary tumor centrally confirmed as triple negative.

Exclusion Criteria:

* locally advanced breast cancers;
* previous breast cancer history;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2591 (Actual)
Dates: Start 2007-12; Primary Completion 2012-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (350):
- United States (43):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Fayetteville, Arkansas
  - Bakersfield, California
  - Fountain Valley, California
  - Greenbrae, California
  - Los Angeles, California
  - Pleasant Hill, California
  - Fairfield, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Orlando, Florida
  - Tamarac, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Lawrenceville, Georgia
  - Niles, Illinois
  - Iowa City, Iowa
  - Waterloo, Iowa
  - Baltimore, Maryland
  - Rockville, Maryland
  - Brownstown, Michigan
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Long Branch, New Jersey
  - The Bronx, New York
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Rutland, Vermont
  - Abingdon, Virginia
  - Richmond, Virginia
- Argentina (2):
  - Buenos Aires
  - Rosario
- Australia (18):
  - Brisbane
  - Camperdown
  - East Bentleigh
  - Fitzroy
  - Geelong
  - Heidelberg
  - Kurralta Park
  - Malvern
  - Nambour
  - Parkville
  - Perth
  - Port Macquarie
  - St Leonards
  - Sydney
  - Wahroonga
  - Waratah
  - Wodonga
  - Wollongong
- Austria (11):
  - Bludesch
  - Graz
  - Innsbruck
  - Krems
  - Leoben
  - Linz
  - Salzburg
  - Vienna
  - Wels
  - Wiener Neustadt
  - Wolfsberg
- Belgium (7):
  - Baudour
  - Brussels
  - Hasselt
  - Namur
  - Sint-Niklaas
  - Tournai
  - Wilrijk
- Sarajevo, Bosnia and Herzegovina
- Brazil (8):
  - Goiânia
  - Ijuí
  - Jaú
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São Paulo
  - Sorocaba
- Canada (20):
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Greater Sudbury, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- China (11):
  - Beijing
  - Changchun
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Shanghai
  - Suzhou
  - Tianjin
  - Wuhan
  - Zhejiang
- San José, Costa Rica
- Czechia (5):
  - Brno
  - Nový Jičín
  - Olomouc
  - Pardubice
  - Prague
- Finland (2):
  - Tampere
  - Turku
- France (26):
  - Angers
  - Bayonne
  - Besançon
  - Bobigny
  - Bordeaux
  - Brest
  - Clermont-Ferrand
  - Colmar
  - Grenoble
  - La Chaussée-Saint-Victor
  - Le Mans
  - Lille
  - Limoges
  - Marseille
  - Montbéliard
  - Montpellier
  - Mougins
  - Nancy
  - Neuilly-sur-Seine
  - Paris
  - Rouen
  - Saint-Cloud
  - Senlis
  - Strasbourg
  - Toulon
  - Tours
- Germany (37):
  - Berlin
  - Bielefeld
  - Bonn
  - Chemnitz
  - Coburg
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Georgsmarienhütte
  - Greifswald
  - Hamburg
  - Heidelberg
  - Herne
  - Kassel
  - Kiel
  - Krefeld
  - Leipzig
  - Lemgo
  - Lüneburg
  - Magdeburg
  - Marburg
  - München
  - Münster
  - Offenbach
  - Offenburg
  - Recklinghausen
  - Rosenheim
  - Stade
  - Trier
  - Tübingen
  - Ulm
  - Weißenfels
  - Wiesbaden
  - Witten
- Greece (3):
  - Heraklion
  - Pátrai
  - Thessaloniki
- Hong Kong, Hong Kong
- Israel (7):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (30):
  - Aviano
  - Bari
  - Bergamo
  - Brescia
  - Brindisi
  - Candiolo
  - Cattolica
  - Cesena
  - Fano
  - Genova
  - Lecce
  - Lido di Camaiore
  - Livorno
  - Lugo
  - Mantova
  - Noale
  - Padua
  - Palermo
  - Parma
  - Pavia
  - Potenza
  - Ravenna
  - Rimini
  - Roma
  - Rozzano
  - San Giovanni Rotondo
  - Sassari
  - Taormina
  - Treviglio
  - Vecchiazzano
- Japan (7):
  - Aichi
  - Ehime
  - Fukuoka
  - Kyoto
  - Osaka
  - Saitama
  - Tokyo
- Malaysia (4):
  - George Town
  - Kelantan
  - Kuala Selangor
  - Petaling Jaya, Selangor
- Mexico (2):
  - León
  - Monterrey
- Netherlands (4):
  - Delftzijl
  - Den Helder
  - Groningen
  - Tilburg
- New Zealand (2):
  - Auckland
  - Wellington
- Skopje, North Macedonia
- Lima, Peru
- Philippines (2):
  - Cebu
  - Quezon City
- Poland (5):
  - Elblag
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
- Portugal (2):
  - Coimbra
  - Lisbon
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (11):
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Moscow
  - Obninsk
  - Persochnysaint-petersburg
  - Ryazan
  - Saint Petersburg
  - Samara
  - Ufa
  - Yekaterinburg
- Serbia (2):
  - Belgrade
  - Kamenitz
- Singapore, Singapore
- South Africa (5):
  - Bloemfontein
  - Durban
  - Johannesburg
  - Pietermaritzburg
  - Pretoria
- South Korea (2):
  - Kyunggi-do
  - Seoul
- Spain (14):
  - Barcelona
  - Burgos
  - Gijón
  - Girona
  - Madrid
  - Mataró
  - Málaga
  - Navarra
  - Palma de Mallorca
  - Pontevedra
  - San Cristóbal de La Laguna
  - Terrassa
  - Valencia
  - Zaragoza
- Sweden (6):
  - Eskilstuna
  - Gävle
  - Lund
  - Malmo
  - Umeå
  - Uppsala
- Switzerland (7):
  - Aarau
  - Basel
  - Bern
  - Chur
  - Thun
  - Winterthur
  - Zurich
- Taiwan (5):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla
- United Kingdom (29):
  - Belfast
  - Birmingham
  - Bournemouth
  - Brighton
  - Bristol
  - Cambridge
  - Cardiff
  - Chelsmford
  - Colchester
  - Dundee
  - Edinburgh
  - Epping
  - Exeter
  - Glasgow
  - Guildford
  - Huddersfield
  - Ipswich
  - Leeds
  - London
  - Manchester
  - Merseyside
  - Newcastle upon Tyne
  - Northwood
  - Peterborough
  - Sheffield
  - Southampton
  - Stoke-on-Trent
  - Truro
  - Wolverhampton

REFERENCES:
- [Derived] Bell R, Brown J, Parmar M, Toi M, Suter T, Steger GG, Pivot X, Mackey J, Jackisch C, Dent R, Hall P, Xu N, Morales L, Provencher L, Hegg R, Vanlemmens L, Kirsch A, Schneeweiss A, Masuda N, Overkamp F, Cameron D. Final efficacy and updated safety results of the randomized phase III BEATRICE trial evaluating adjuvant bevacizumab-containing therapy in triple-negative early breast cancer. Ann Oncol. 2017 Apr 1;28(4):754-760. doi: 10.1093/annonc/mdw665. PMID 27993816
- [Derived] Cameron D, Brown J, Dent R, Jackisch C, Mackey J, Pivot X, Steger GG, Suter TM, Toi M, Parmar M, Laeufle R, Im YH, Romieu G, Harvey V, Lipatov O, Pienkowski T, Cottu P, Chan A, Im SA, Hall PS, Bubuteishvili-Pacaud L, Henschel V, Deurloo RJ, Pallaud C, Bell R. Adjuvant bevacizumab-containing therapy in triple-negative breast cancer (BEATRICE): primary results of a randomised, phase 3 trial. Lancet Oncol. 2013 Sep;14(10):933-42. doi: 10.1016/S1470-2045(13)70335-8. Epub 2013 Aug 7. PMID 23932548

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab and Chemotherapy: Participants randomized to receive bevacizumab and chemotherapy.
  For these patients, bevacizumab was given in combination with chemotherapy at a dose of 5 mg/kg/week equivalent using 1 of 3 different scheduling options depending on the schedule of the adjuvant chemotherapy selected. After completing chemotherapy + bevacizumab (treatment period 1), patients in this arm received bevacizumab monotherapy up to a total duration of 1 year (treatment period 2).
  At the end of treatment (i.e., after approximately 55 weeks), patients were followed up until the end of the study.
- Chemotherapy: Participants randomized to receive chemotherapy alone.
  For patients randomized to the chemotherapy alone arm, investigators could select from one of three chemotherapy regimens. After completing chemotherapy (treatment period 1) patients entered a post-treatment surveillance period for the remainder of the first year after randomization (treatment period 2).
  At the end of treatment (i.e., after approximately 55 weeks), patients were followed up until the end of the study.
Period: Overall Study
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Started | 1301 | 1290
Intention to Treat | 1301 | 1290
Safety Population | 1288 | 1271
Completed | 870 | 982
Not Completed | 431 | 308
Not completed — Death | 4 | 5
Not completed — Breast Cancer Recurrence/2nd Primary | 30 | 60
Not completed — Adverse Event/Intermittent Illness | 255 | 29
Not completed — Violation Criteria at Entry | 3 | 17
Not completed — Withdrew Consent | 59 | 55
Not completed — Refused Treatment/Did Not Cooperate | 52 | 42
Not completed — Failure to Return | 1 | 4
Not completed — Other Protocol Violation | 5 | 21
Not completed — Administrative/Other | 22 | 75

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab and Chemotherapy: Participants randomized to receive bevacizumab and chemotherapy
- Chemotherapy: Participants randomized to receive chemotherapy alone
- Total: Total of all reporting groups
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy | Total
Number analyzed (Participants) | 1301 | 1290 | 2591
Age, Customized [Number; unit: participants]
  < 40 years | 231 | 253 | 484
  >= 40 to < 65 years | 952 | 916 | 1868
  >= 65 years | 118 | 121 | 239
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1301 | 1290 | 2591
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Invasive Disease-free Survival (IDFS) Event
Description: IDFS, was a composite endpoint defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site);Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer or Second primary non-breast invasive cancer.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.1810, Log Rank; Stratification factors were axillary nodal status, choice of adjuvant chemotherapy, hormone receptor status, surgery; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.07]

2. Secondary Outcome: Time to Overall Survival (OS) Event
Description: OS was defined as the time from randomization to death attributable to any cause. Patients for whom no death is captured in the clinical database up to the clinical cut-off date are censored at the last time they were known to be alive.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Chemotherapy: Participants randomized to receive chemotherapy
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached | NA [NA to NA] — The median was not reached

3. Secondary Outcome: Time to Overall Survival (OS) Event
Description: as for outcome 2
Time Frame: Event driven (until data cutoff: 30 June 2014: up to 77 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not estimable. | NA [NA to NA] — The median was not estimable.
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.5247, Log Rank; Stratification factors are Axillary nodal status, Choice of adjuvant chemotherapy, Hormone receptor status, Surgery; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.74 to 1.17]

4. Primary Outcome: Percentage of Participants With Invasive Disease-free Survival (IDFS) Events
Description: IDFS, was a composite endpoint defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site);Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer or Second primary non-breast invasive cancer. The percentage of participants with and without IDFS Events by the time of the data cutoff is presented.
Time Frame: Event driven (until data cutoff: 29 February 2012 up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Percentage of participants
  Percentage of Participants with Events | 14.5 | 15.9
  Percentage of Participants without Events | 85.5 | 84.1

5. Primary Outcome: Time to Invasive Disease-free Survival (IDFS) Event Excluding Second Primary Non-Breast Invasive Cancer
Description: IDFS, was a composite endpoint defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site); Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.1966, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.07] — Stratification factors were axillary nodal status, choice of adjuvant chemotherapy, hormone receptor status, surgery

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS) Event
Description: as for outcome 2
Time Frame: Event driven (until data cut off: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
percentage of participants
  with events | 7.1 | 8.3
  without events | 92.9 | 91.7
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.2318, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.12]

7. Primary Outcome: Percentage of Participants With Invasive Disease-free Survival (IDFS) Events Excluding Second Primary Non-Breast Invasive Cancer
Description: IDFS, was a composite endpoint defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site); Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer. Percentage of participants with and without IDFS Events by the time of data cutoff is presented.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Percentage of participants
  Percentage of Participants with Events | 13.5 | 14.7
  Percentage of Participants without Events | 86.5 | 85.3

8. Secondary Outcome: Percentage of Participants With Overall Survival (OS) Event
Description: as for outcome 2
Time Frame: Event driven (until data cut off: 30 June 2014: up to 77 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
percentage of participants
  with events | 11.1 | 11.6
  without events | 88.9 | 88.4

9. Secondary Outcome: Time to Breast Cancer-Free Interval (BCFI) Event
Description: BCFI is defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral local/regional invasive breast cancer recurrence or distant breast cancer recurrence; Contralateral invasive breast cancer; Ipsilateral or contralateral Ductal carcinoma in situ or Death only from breast cancer cause.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat participants, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.2792, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.72 to 1.10] — Stratification factors were axillary nodal status, choice of adjuvant chemotherapy, hormone receptor status, surgery

10. Secondary Outcome: Percentage of Participants With Breast Cancer-Free Interval (BCFI) Events
Description: BCFI is defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral local/regional invasive breast cancer recurrence or distant breast cancer recurrence; Contralateral invasive breast cancer; Ipsilateral or contralateral DCIS or Death only from breast cancer cause. Percentage of participants with and without BCFI events by the time of the data cutoff is presented.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Percentage of participants
  Percentage of Participants with Events | 13.2 | 14.2
  Percentage of Participants without Events | 86.8 | 85.8

11. Secondary Outcome: Time to Disease-Free Survival (DFS) Event
Description: DFS is defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site); Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer, Second primary non-breast invasive cancer or New diagnosis of an ipsilateral or contralateral Ductal carcinoma in situ (DCIS).
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.1832, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.07] — Stratification factors were axillary nodal status, choice of adjuvant chemotherapy, hormone receptor status, surgery

12. Secondary Outcome: Percentage of Participants With Disease-Free Survival (DFS) Events
Description: DFS is defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast cancer recurrence (same breast); Ipsilateral (same side of body) local regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and/or skin); Distant recurrence (evidence of breast cancer in any anatomic site); Death attributable to any cause; Contralateral (opposite side of the body) invasive breast cancer, Second primary non-breast invasive cancer or New diagnosis of an ipsilateral or contralateral Ductal carcinoma in situ (DCIS). Percentage of Participants with and without DFI Events by the time of the data cut-off is presented.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Percentage of participants
  with Events | 14.7 | 16.1
  without Events | 85.3 | 83.9

13. Secondary Outcome: Time to Distant Disease-Free Survival (DDFS) Event
Description: DDFS is defined as the time from randomization until the date of the first occurrence of one of the following events: Distant recurrence; Death attributable to any cause; Second primary non-breast invasive cancer (with the exception of non-melanoma Skin cancers).
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached
Statistical Analysis 1: Comparison: Bevacizumab and Chemotherapy vs Chemotherapy; Test type: Superiority or Other; p = 0.3309, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.12] — Stratification factors were axillary nodal status, choice of adjuvant chemotherapy, hormone receptor status, surgery

14. Secondary Outcome: Percentage of Participants With Distant Disease-Free Survival (DDFS) Events
Description: DDFS is defined as the time from randomization until the date of the first occurrence of one of the following events: Distant recurrence; Death attributable to any cause; Second primary non-breast invasive cancer (with the exception of non-melanoma Skin cancers). Percentage of participants with and without DDFS Events by the time of the data cutoff is presented.
Time Frame: Event driven (until data cutoff: 29 February 2012: up to 49 months)
Population: Intent-to-treat population, defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab and Chemotherapy | Chemotherapy
Number analyzed (Participants) | 1301 | 1290
Percentage of participants
  Percentage of Participants with Events | 11.7 | 12.7
  Percentage of Participants without Events | 88.3 | 87.3

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) and Deaths
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is Life-Threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Through end of study: 30 June 2014: up to 77 months
Population: Safety population, defined as all randomized participants who received at least one dose of study drug. Participants who received at least one full or partial dose of bevacizumab were included in the bevacizumab and chemotherapy arm; all other patients were analyzed in the chemotherapy arm.
Measure: Number; unit: Participants
Groups:
- Bevacizumab and Chemotherapy (0-18 Months): Occurring in participants who received bevacizumab and chemotherapy, 0-18 months after first dose
- Chemotherapy (0-18 Months): Occurring in participants who received chemotherapy alone, 0-18 months after first dose
- Bevacizumab and Chemotherapy (>18 Months): Occurring in participants who received bevacizumab and chemotherapy, more than 18 months after first dose
- Chemotherapy (>18 Months): Occurring in participants who received chemotherapy alone, more than 18 months after first dose
Arm/Group | Bevacizumab and Chemotherapy (0-18 Months) | Chemotherapy (0-18 Months) | Bevacizumab and Chemotherapy (>18 Months) | Chemotherapy (>18 Months)
Number analyzed (Participants) | 1288 | 1271 | 1288 | 1271
Participants
  Serious Adverse Events | 379 | 250 | 45 | 48
  Adverse Events (5% Reporting Threshold) | 1268 | 1233 | 0 | 0
  Deaths | 31 | 41 | 113 | 106

ADVERSE EVENTS:
Time Frame: Through end of study, 30 June 2014
Description: The analysis set was the safety population, defined as all randomized participants who received at least one dose of study drug. Participants who received at least one full or partial dose of bevacizumab were included in the bevacizumab and chemotherapy arm; all others, in the chemotherapy arm. MedDRA (15.0) and MedDRA (17.0) were used.
Groups:
- Bevacizumab and Chemotherapy (0-18 Months): Occurring in participants who received bevacizumab and chemotherapy, during treatment period (0-18 months) after first dose
- Chemotherapy (0-18 Months): Occurring in participants who received chemotherapy alone, during treatment period (0-18 months) after first dose
- Bevacizumab and Chemotherapy (>18 Months): Occurring in participants who received bevacizumab and chemotherapy, during follow-up period (>18 months) after first dose
- Chemotherapy (>18 Months): Occurring in participants who received chemotherapy alone, during follow-up period (>18 months) after first dose
Arm/Group | Bevacizumab and Chemotherapy (0-18 Months) | Chemotherapy (0-18 Months) | Bevacizumab and Chemotherapy (>18 Months) | Chemotherapy (>18 Months)
Serious Adverse Events (participants affected / at risk) | 379/1288 | 250/1271 | 45/1288 | 48/1271
Other Adverse Events (participants affected / at risk) | 1268/1288 | 1233/1271 | 0/1288 | 0/1271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Chemotherapy (0-18 Months) (N=1288) | Chemotherapy (0-18 Months) (N=1271) | Bevacizumab and Chemotherapy (>18 Months) (N=1288) | Chemotherapy (>18 Months) (N=1271)
Febrile neutropenia (Blood and lymphatic system disorders) | 84 | 59 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 69 | 38 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 13 | 11 | 0 | 0
Infection (Infections and infestations) | 14 | 3 | 0 | 1
Device related infection (Infections and infestations) | 9 | 4 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 6 | 0 | 0
Neutropenic infection (Infections and infestations) | 8 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 4 | 5 | 0 | 1
Cellulitis (Infections and infestations) | 5 | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 0 | 1
Anal abscess (Infections and infestations) | 5 | 0 | 0 | 0
Sepsis (Infections and infestations) | 4 | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 3 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 3 | 0 | 0
Mastitis (Infections and infestations) | 2 | 2 | 2 | 1
Wound infection (Infections and infestations) | 3 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 2 | 0 | 0
Breast cellulitis (Infections and infestations) | 1 | 1 | 1 | 2
Febrile infection (Infections and infestations) | 2 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0 | 0 | 0
Breast infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0
Lymph node abscess (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 9 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 12 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 4 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Enterocolonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 21 | 19 | 0 | 0
General physical health deterioration (General disorders) | 5 | 2 | 0 | 0
Chest pain (General disorders) | 3 | 3 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 2 | 0 | 0
Thrombosis in device (General disorders) | 2 | 1 | 0 | 0
Device damage (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Patient-device incompatibility (General disorders) | 2 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Device deployment issue (General disorders) | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 1 | 0 | 0 | 0
Device extrusion (General disorders) | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 6 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 4 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 5 | 0 | 1
Hypertension (Vascular disorders) | 7 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 5 | 2 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 7 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0
Cytology abnormal (Investigations) | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
IGA nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 2 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Gaze palsy (Eye disorders) | 0 | 0 | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lipogranuloma (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Rehabilitation therapy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Antiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast calcifications (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Chemotherapy (0-18 Months) (N=1288) | Chemotherapy (0-18 Months) (N=1271) | Bevacizumab and Chemotherapy (>18 Months) (N=1288) | Chemotherapy (>18 Months) (N=1271)
Nausea (Gastrointestinal disorders) | 881 | 880 |  |
Stomatitis (Gastrointestinal disorders) | 663 | 469 |  |
Vomiting (Gastrointestinal disorders) | 480 | 459 |  |
Constipation (Gastrointestinal disorders) | 444 | 401 |  |
Diarrhoea (Gastrointestinal disorders) | 418 | 350 |  |
Dyspepsia (Gastrointestinal disorders) | 201 | 165 |  |
Abdominal pain upper (Gastrointestinal disorders) | 138 | 112 |  |
Abdominal pain (Gastrointestinal disorders) | 123 | 124 |  |
Gingival bleeding (Gastrointestinal disorders) | 138 | 10 |  |
Dry mouth (Gastrointestinal disorders) | 61 | 76 |  |
Haemorrhoids (Gastrointestinal disorders) | 78 | 58 |  |
Alopecia (Skin and subcutaneous tissue disorders) | 807 | 833 |  |
Nail disorder (Skin and subcutaneous tissue disorders) | 183 | 150 |  |
Rash (Skin and subcutaneous tissue disorders) | 160 | 137 |  |
Erythema (Skin and subcutaneous tissue disorders) | 86 | 114 |  |
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 92 | 70 |  |
Dry skin (Skin and subcutaneous tissue disorders) | 70 | 72 |  |
Pruritus (Skin and subcutaneous tissue disorders) | 71 | 63 |  |
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 68 | 49 |  |
Fatigue (General disorders) | 533 | 539 |  |
Asthenia (General disorders) | 230 | 223 |  |
Pyrexia (General disorders) | 214 | 164 |  |
Oedema peripheral (General disorders) | 145 | 164 |  |
Pain (General disorders) | 72 | 58 |  |
Influenza like illness (General disorders) | 68 | 61 |  |
Arthralgia (Musculoskeletal and connective tissue disorders) | 414 | 252 |  |
Myalgia (Musculoskeletal and connective tissue disorders) | 278 | 273 |  |
Pain in extremity (Musculoskeletal and connective tissue disorders) | 198 | 171 |  |
Back pain (Musculoskeletal and connective tissue disorders) | 172 | 141 |  |
Bone pain (Musculoskeletal and connective tissue disorders) | 99 | 111 |  |
Headache (Nervous system disorders) | 440 | 289 |  |
Dysgeusia (Nervous system disorders) | 243 | 230 |  |
Neuropathy peripheral (Nervous system disorders) | 138 | 135 |  |
Peripheral sensory neuropathy (Nervous system disorders) | 137 | 128 |  |
Dizziness (Nervous system disorders) | 130 | 121 |  |
Paraesthesia (Nervous system disorders) | 88 | 91 |  |
Neutropenia (Blood and lymphatic system disorders) | 503 | 479 |  |
Leukopenia (Blood and lymphatic system disorders) | 210 | 215 |  |
Anaemia (Blood and lymphatic system disorders) | 140 | 175 |  |
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 478 | 75 |  |
Cough (Respiratory, thoracic and mediastinal disorders) | 215 | 161 |  |
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 179 | 99 |  |
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 144 | 123 |  |
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 104 | 65 |  |
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 99 | 19 |  |
Hypertension (Vascular disorders) | 456 | 65 |  |
Hot flush (Vascular disorders) | 206 | 208 |  |
Lymphoedema (Vascular disorders) | 70 | 74 |  |
Nasopharyngitis (Infections and infestations) | 137 | 125 |  |
Upper respiratory tract infection (Infections and infestations) | 103 | 109 |  |
Urinary tract infection (Infections and infestations) | 95 | 100 |  |
Insomnia (Psychiatric disorders) | 191 | 217 |  |
Anxiety (Psychiatric disorders) | 88 | 78 |  |
Depression (Psychiatric disorders) | 57 | 69 |  |
Decreased appetite (Metabolism and nutrition disorders) | 260 | 223 |  |
Ejection fraction decreased (Investigations) | 103 | 71 |  |
Aspartate aminotransferase increased (Investigations) | 84 | 49 |  |
Gamma-glutamyltransferase increased (Investigations) | 82 | 45 |  |
Alanine aminotransferase increased (Investigations) | 67 | 50 |  |
Weight decreased (Investigations) | 72 | 28 |  |
Left ventricular dysfunction (Cardiac disorders) | 261 | 165 |  |
Radiation skin injury (Injury, poisoning and procedural complications) | 151 | 190 |  |
Lacrimation increased (Eye disorders) | 156 | 109 |  |
Proteinuria (Renal and urinary disorders) | 195 | 24 |  |
Breast pain (Reproductive system and breast disorders) | 60 | 86 |  |
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 162 | 123 |  |

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.